CLINICAL TRIAL: NCT03248167
Title: Cannabidiol as a Treatment for Alcohol Use Disorder Comorbid With Posttraumatic Stress Disorder
Brief Title: Cannabidiol as a Treatment for AUD Comorbid With PTSD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Tilray (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00949
Record Dates: First submitted 2017-08-02; First posted 2017-08-14 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
Keywords: Cannabidiol
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD 600 mg daily) (Experimental): 6 weeks, such that both participants and study staff are blind to treatment condition.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): 6 weeks, such that both participants and study staff are blind to treatment condition.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Cannabidiol — 600 mg daily
  Other Names: CBD
  Arms: Cannabidiol (CBD 600 mg daily)
Drug: Placebos — This project aims to determine whether cannabidiol (CBD) is effective in treating alcohol use disorder (AUD) comorbid posttraumatic stress disorder (PTSD). To address this aim, investigators will conduct a clinical trial in which CBD will be administered to 48 individuals with AUD comorbid with PTSD, and assess alcohol intake and PTSD symptoms. The aim is to test the hypothesis that CBD will reduce alcohol drinking in individuals with AUD comorbid with PTSD. To test this hypothesis, 48 otherwise healthy adult participants with moderate or severe AUD and PTSD will be randomized to treatment with either CBD (600 mg daily) or placebo, for a period of 6 weeks, such that both participants and study staff are blind to treatment condition.
  Arms: Placebo

SUMMARY:
This project aims to determine whether cannabidiol (CBD), a compound derived from the cannabis plant, is effective in treating alcohol use disorder (AUD) in individuals with comorbid posttraumatic stress disorder (PTSD). Investigators will test the hypothesis that oral cannabidiol (CBD) will reduce alcohol drinking in individuals with AUD comorbid with PTSD. To test this hypothesis, 48 otherwise healthy adult participants with moderate or severe AUD and PTSD will be randomized to treatment with either CBD (600 mg daily) or placebo, for a period of 6 weeks, such that both participants and study staff are blind to treatment condition. Participants (each treated for 6 weeks) will be continuously recruited over a study period of 14 months until 48 have completed. Baseline and weekly data will be collected on alcohol usage and PTSD symptoms, and investigators will assess whether CBD treatment leads to a greater improvement in these measures relative to placebo, and whether reduction in alcohol drinking is temporally linked to improvement in PTSD symptoms. Subjects will also participate in a task designed to quantify the psychological and physiological links between negative emotion produced by re-experiencing PTSD trauma, and alcohol craving. The task will be administered following 4 weeks of treatment. Treatment-associated reduction in alcohol craving elicited by trauma-associated negative emotion between CBD and placebo groups will be compared. This study will be the first to test whether CBD is effective in treating alcohol addiction and in treating PTSD in humans, and the first to examine the interaction between these treatment effects. Results will serve as proof of concept and provide guidance for a future larger clinical trial. Because CBD is a safe, readily available drug, such a trial would have an immense potential to prevent death, medical illness, and psychological suffering associated with AUD and PTSD. Further, because the brain circuits via which CBD acts to produce hypothesized effects are relatively well-understood, results may substantially advance understanding of the neurobiological basis of alcohol addiction.

DETAILED DESCRIPTION:
In this project, investigators aim to test the hypothesis that CBD will reduce alcohol drinking in individuals with AUD comorbid with PTSD. CBD is currently a medical research focus because it shows promise for treating anxiety and other brain disorders, but does not produce a 'high' like other parts of cannabis, has not been shown to be addictive, and is safe, with few or no side effects. AUD, which is one of the most common and most debilitating psychiatric conditions, is often associated with other comorbid psychiatric disorders - in particular, PTSD: depending on the population studied, 30-60% of individuals with AUD also have PTSD, with high comorbidity rates in military veterans. Evidence from animal models and clinical studies suggests that the negative emotion caused by PTSD symptoms intensifies craving for alcohol during alcohol withdrawal, perpetuating the addictive cycle; further, evidence shows that the brain circuits underlying negative emotion and addiction are linked in a forebrain area called the extended amygdala, which provides a neuropharmacological target to simultaneously treat both negative emotion and alcohol addiction in individuals with AUD and PTSD. CBD is known to inhibit brain activity in the extended amygdala, leading to reduced anxiety in both animal models and humans. CBD also reduces addictive alcohol seeking in animal models.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-70
2. DSM-5 diagnosis of moderate or severe AUD
3. DSM-5 diagnosis of PTSD with Clinician Administered PTSD Scale (CAPS-5) OR subPTSD diagnosis (meeting criterion A, F, G, H and at least 6 symptoms across any criteria B-E) with Clinician Administered PTSD Scale (CAPS-5)
4. Able to provide voluntary informed consent
5. At least 6 heavy drinking days (4 or more drinks per day for a woman, 5 or more drinks per day for a man) in the 30 days prior to screen
6. If of childbearing potential (male or female), are willing to use approved form of contraception from screening for duration of the trial
7. Able to provide at least two locators
8. Endorse desire to cut down or stop drinking
9. Agrees to abstain from all other cannabinoid use for the duration of the study
10. Confirms they are reliably domiciled

Exclusion Criteria:

1. Current alcohol withdrawal (CIWA-Ar score >7)
2. Exclusionary medical conditions (e.g. current severe alcohol withdrawal requiring medical hospitalization, significantly impaired liver function)
3. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder
4. High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process, based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support)
5. Exposure to trauma in the last 30 days, including police duty or military service
6. Current significant suicidality (assessed using the C-SSRS), any significant suicidal behavior in the past 12 months, or any history of serious suicide attempts requiring hospitalization, or current significant homicidality
7. History of Severe Traumatic Brain Injury (TBI; as indicated by Loss of Consciousness > 24 hours)
8. DSM-5 diagnosis of current mild cannabis use disorder and/or moderate or severe substance use disorder for a substance other than alcohol or nicotine
9. Significant laboratory abnormalities, including significantly impaired liver function, serious abnormalities of complete blood count or metabolic panel
10. Active legal problems likely to result in incarceration within 12 weeks of treatment initiation
11. Pregnancy or lactation
12. Current use of exclusionary medications, including but not limited to cannabinoids; those acting on serotonergic pathways; treatments for addictions including alcohol; moderate to strong inhibitors of CYP3A4 or CYP2C19; medications metabolized primarily by CYP3A4, CYP3A5, or CYP3A7; and medications with a narrow therapeutic index which are substrates of UGT1A9, UGT2B7, CYP2C8, CYP2C9, CYP2C19, CYP1A2, or CYP2B6.
13. Current treatment for AUD (with exceptions of: AA/12-step treatment and/or psychosocial treatment initiated more than 3 months prior to the screening visit)
14. Psychotherapy for PTSD or other psychiatric condition, if initiated within 3 months of screening
15. Inpatient psychiatric treatment in the last 12 months, with the exception of detox and extended Emergency Department stays
16. A positive urine drug screen for opioids at screen, baseline, or any later visits. If a participant has a positive drug screen for THC or cocaine at screen, baseline or a later visit- their enrollment will be subject to the clinical judgement of the Principal Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 95 patients were enrolled in the trial. 65 of those failed screening or were lost to follow-up prior to starting medication. Thus, only 30 participants started medication in the trial.
Groups:
- Placebo: 6 weeks, such that both participants and study staff are blind to treatment condition.
  Placebos: This project aims to determine whether cannabidiol (CBD) is effective in treating alcohol use disorder (AUD) comorbid posttraumatic stress disorder (PTSD). To address this aim, investigators will conduct a clinical trial in which CBD will be adminstred to 48 individuals with AUD comorbid with PTSD, and assess alcohol intake and PTSD symptoms. The aim is to test the hypothesis that CBD will reduce alcohol drinking in individuals with AUD comorbid with PTSD. To test this hypothesis, 48 otherwise healthy adult participants with moderate or severe AUD and PTSD will be randomized to treatment with either CBD (600 mg daily) or placebo, for a period of 6 weeks, such that both participants and study staff are blind to treatment condition.
Period: Overall Study
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Started | 17 | 13
Completed | 12 | 9
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Institution Mandated COVID-19 Research Pause | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Full Range); unit: years] | 38.59 [22 to 61] | 37.69 [21 to 54] | 38.2 [21 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 7 | 7 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Per Day
Description: Number of drinks per day will be assessed by the Time Line Follow Back (TLFB) methodology. TLFB is a drinking assessment method that can be administered in various formats: as clinician-administered interview, paper and pencil and computer. TLFB is used to obtain estimates of the quantity of daily drinking.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: drinks/day
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
drinks/day | 4.4885 (2.6620) | 5.3623 (2.7075)

2. Primary Outcome: Number of Drinks Per Day
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: drinks/day
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 10
drinks/day | 1.9256 (2.1786) | 2.15 (2.2792)

3. Primary Outcome: Number of Drinks Per Day
Description: as for outcome 1
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: drinks/day
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
drinks/day | 2.4881 (2.1679) | 2.8175 (2.2682)

4. Primary Outcome: PCL-5 Total Score
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of post-traumatic stress disorder (PTSD). The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; the higher the score, the more severe the PTSD symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
score on a scale | 42.0588 (13.8549) | 49.1538 (13.7739)

5. Primary Outcome: PCL-5 Total Score
Description: as for outcome 4
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 13 | 10
score on a scale | 19.9231 (15.7116) | 29.9 (16.7559)

6. Primary Outcome: PCL-5 Total Score
Description: as for outcome 4
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 11 | 9
score on a scale | 26.6364 (18.4921) | 26.8889 (17.7331)

7. Secondary Outcome: Percent Carbohydrate Deficient Transferrin (CDT)
Description: CDT test performed on blood sample
Time Frame: Baseline
Measure: Mean (Full Range); unit: percentage of CDT
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
percentage of CDT | 1.1118 [0.6 to 2.6] | 2.2833 [0.5 to 8.8]

8. Secondary Outcome: Percent Carbohydrate Deficient Transferrin (CDT)
Description: CDT test performed on blood sample
Time Frame: Week 4
Measure: Mean (Full Range); unit: percentage of CDT
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 11 | 9
percentage of CDT | 1.0909 [0.6 to 2.1] | 1.4222 [0.6 to 3.4]

9. Secondary Outcome: Percent Carbohydrate Deficient Transferrin (CDT)
Description: CDT test performed on blood sample
Time Frame: Week 6
Measure: Mean (Full Range); unit: percentage of CDT
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 10 | 8
percentage of CDT | 1.14 [0.7 to 1.9] | 1.6625 [0.6 to 5.8]

10. Secondary Outcome: Percentage of Heavy Drinking Days
Description: Heavy drinking days is defined as 4+ drinks for women or five or more drinks for men per drinking day. This will be averaged for each treatment week.
Time Frame: Baseline
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
percentage of days | 49 [17 to 97] | 58 [13 to 100]

11. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 1
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 13
percentage of days | 29 [0 to 100] | 31 [0 to 100]

12. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 2
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 12
percentage of days | 25 [0 to 100] | 31 [0 to 100]

13. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 3
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 14 | 11
percentage of days | 21 [0 to 100] | 21 [0 to 100]

14. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 4
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 23 [0 to 100] | 25 [0 to 100]

15. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 5
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 26 [0 to 100] | 32 [0 to 86]

16. Secondary Outcome: Percentage of Heavy Drinking Days
Description: as for outcome 10
Time Frame: Week 6
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 21 [0 to 100] | 39 [0 to 100]

17. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: Very heavy drinking days is defined as 8+/10+ drinks per day for women and men respectively. This will be averaged for each treatment week.
Time Frame: Baseline
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
percentage of days | 17 [0 to 67] | 27 [0 to 77]

18. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 1
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
percentage of days | 4 [0 to 25] | 4 [0 to 25]

19. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 2
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 12
percentage of days | 4 [0 to 29] | 4 [0 to 33]

20. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 3
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 14 | 11
percentage of days | 5 [0 to 43] | 1 [0 to 14]

21. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 4
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 10
percentage of days | 1 [0 to 14] | 1 [0 to 14]

22. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 5
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 2 [0 to 14] | 3 [0 to 29]

23. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: as for outcome 17
Time Frame: Week 6
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 2 [0 to 14] | 5 [0 to 29]

24. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
Participants | 5 | 4

26. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 12
Participants | 6 | 6

27. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 14 | 11
Participants | 9 | 6

28. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 10
Participants | 7 | 5

29. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
Participants | 5 | 5

30. Secondary Outcome: Number of Participants With No Heavy Drinking Days
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
Participants | 4 | 4

31. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
Participants | 17 | 13

32. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 13
Participants | 16 | 13

33. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 13
Participants | 16 | 13

34. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 14 | 11
Participants | 14 | 11

35. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 10
Participants | 12 | 10

36. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
Participants | 12 | 9

37. Secondary Outcome: Number of Participants That Are 'Present and Clear'
Description: Present is defined as present to provide breath alcohol levels (BAC). Clear is defined as having a BAC of zero.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
Participants | 12 | 9

38. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Baseline
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 17 | 13
percentage of days | 30 [0 to 77] | 34 [0 to 87]

39. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 1
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 13
percentage of days | 55 [0 to 100] | 57 [0 to 100]

40. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 2
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 16 | 13
percentage of days | 55 [0 to 100] | 53 [0 to 100]

41. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 3
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 14 | 11
percentage of days | 66 [0 to 100] | 56 [0 to 100]

42. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 4
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 10
percentage of days | 56 [0 to 100] | 57 [0 to 100]

43. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 5
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 52 [0 to 100] | 51 [0 to 100]

44. Secondary Outcome: Percentage of Days Abstinent
Time Frame: Week 6
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
Number analyzed (Participants) | 12 | 9
percentage of days | 48 [0 to 100] | 46 [0 to 100]

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Collection approach was systematic, a study Nurse Practitioner of Physician collected the SAFTEE form Part A (with Parts B and C as needed) to collect AEs from a list of known drug effects. This assessment includes questions related to description of AE, timeline, severity, relatedness to study drug/participation, etc. This assessment was completed on a weekly basis from the baseline assessment to week 7 and then again at the week 9 followup. All AEs were reviewed with the PI.
Arm/Group | Cannabidiol (CBD 600 mg Daily) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 15/17 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (CBD 600 mg Daily) (N=17) | Placebo (N=13)
Anxiety (Psychiatric disorders) | 0 | 1
Lightheadedness/Dizziness (General disorders) | 1 | 1
Thyroid Nodule (Endocrine disorders) | 1 | 0
Acid Reflux (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurry Vision (Eye disorders) | 1 | 1
Cold/Flu Symptoms (General disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Drowsiness (General disorders) | 6 | 4
Elevated liver enzymes (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Feeling Overwhelmed (Psychiatric disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Headache (Gastrointestinal disorders) | 2 | 0
Hypotension (Cardiac disorders) | 1 | 0
Increased Hunger (General disorders) | 2 | 1
Insomnia (General disorders) | 1 | 1
Irregular heartbeat (Cardiac disorders) | 0 | 1
Lack of motivation (Psychiatric disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Nightmares (General disorders) | 1 | 2
Perceptual problems (General disorders) | 1 | 0
Arm surgery (Musculoskeletal and connective tissue disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Weight gain (General disorders) | 3 | 2
Shortness of breath (Vascular disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 1
Suicidal ideation (wish to be dead) (Psychiatric disorders) | 1 | 0
Sweating (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03248167/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03248167/ICF_000.pdf